CLINICAL TRIAL: NCT05827484
Title: A New Treatment Modality For Skeletal Muscles Sports Injuries; Losartan Combination With PRP
Brief Title: The Effect of Combined Use of Anti-fibrotic Agent With Platelet Rich Plasma on Skeletal Muscle Healing After Acute Injuries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mostafa Hassanein, Msc (Other)
Responsible Party: Sponsor-Investigator, Mostafa Hassanein, Msc, principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MS 22/2016
Record Dates: First submitted 2023-04-01; First posted 2023-04-25 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: PRP; Losartan; Muscle Injury; Sport Injury
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10 patients with acute skeletal muscle injury underwent PRP injection (Active Comparator): Patients with acute skeletal muscle injury received a single ultrasound guided local PRP injection in the site of injury in day 1 or 2 of the injury.
  Interventions: Biological: Autologous platelets rich plasma
- 10 patients with acute skeletal muscle injury underwent PRP injection and oral LOSARTAN (Experimental): Patients with acute skeletal muscle injury received a single ultrasound guided local PRP injection in day 1 or 2 of injury in addition to administration of oral (50mg LOSARTAN /day) from day 5 to day 30.
  Interventions: Combination Product: Autologous platelets rich plasma + oral LOSARTAN administration

INTERVENTIONS:
Biological: Autologous platelets rich plasma — 30 ml of venous blood were drawn from the participant by means of venipuncture. The collected blood was mixed with 3 ml anti-coagulant acid citrate dextrose in the centrifugation sterile tube. The blood sample was then centrifuged using the centrifugation machine. 3 ml of PRP from the buffy coat layer were loaded in a 5 ml syringe. After local sterilization and draping of the site of injection and under US guidance the hematoma was aspirated from the injury site and the freshly prepared PRP was injected.
  Other Names: PRP
  Arms: 10 patients with acute skeletal muscle injury underwent PRP injection
Combination Product: Autologous platelets rich plasma + oral LOSARTAN administration — in addition to local PRP injection, 50 mg / day of LOSARTAN (Cozaar® 50 mg film-coated tablets) were administrated to the study group orally every morning from day 5 and till day 30 after injury.
  Other Names: PRP + LOSARTAN
  Arms: 10 patients with acute skeletal muscle injury underwent PRP injection and oral LOSARTAN

SUMMARY:
The aim of this comparative study is to determine whether or not LOSARTAN with its anti-fibrotic action has an added effect when administrated with platelet rich plasma injection on skeletal muscle healing and on decreasing the fibrous scar after muscle injuries in comparison with the sole administration of platelet rich plasma.

ELIGIBILITY:
Inclusion Criteria:

* Adult age. (18 - 40 year old).
* Clinically diagnosed acute skeletal muscle injury with maximum 3 days duration and ultrasonographically confirmed grade II according to Woodhouse et al.
* Understanding the study and accepting the participation

Exclusion Criteria:

* Any connective tissue disease (e.g. rheumatoid arthritis, systemic lupus erythematous, etc.)
* Hypertension or hypotension
* Diabetes mellitus
* Any cardiac or pulmonary disease
* NSAIDs use in less than a week prior to the beginning of the study.
* Muscle injuries requiring surgical interference.
* No detectable injury ultrasonographically.
* Anemia
* Thrombocytopenia or any platelet disorder.
* Pregnancy or lactation.
* Local infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
ecchymosis | 1or 2 days after injury
  locally at the site of injury "present or absent"
ecchymosis | 2 weeks after injury.
  locally at the site of injury "present or absent"
ecchymosis | 1month after injury.
  locally at the site of injury "present or absent"
ecchymosis | 3 months after injury.
  locally at the site of injury "present or absent"
deformity | 1 or 2 days after injury
  palpable defects at the site of injury "present or absent"
deformity | 2 weeks after injury.
  palpable defects at the site of injury "present or absent"
deformity | 1month after injury.
  palpable defects at the site of injury "present or absent"
deformity | 3 months after injury.
  palpable defects at the site of injury "present or absent"
tenderness | 1 or 2 days after injury
  at the site of injury "present or absent"
tenderness | 2 weeks after injury.
  at the site of injury "present or absent"
tenderness | 1month after injury.
  at the site of injury "present or absent"
tenderness | 3 months after injury.
  at the site of injury "present or absent"
Pain at site of injury | 1 or 2 days after injury
  pain at site of injury using visual analog score "VAS" where 0 is lowest and 100 is highest pain
Pain at site of injury | 2 weeks after injury.
  pain at site of injury using visual analog score "VAS" where 0 is lowest and 100 is highest pain
Pain at site of injury | 1month after injury.
  pain at site of injury using visual analog score "VAS" where 0 is lowest and 100 is highest pain
Pain at site of injury | 3 months after injury.
  pain at site of injury using visual analog score "VAS" where 0 is lowest and 100 is highest pain
spasm | 1or 2 days after injury.
  spasm in the injured muscle "present or absent"
spasm | 2 weeks after injury.
  spasm in the injured muscle "present or absent"
spasm | 1month after injury.
  spasm in the injured muscle "present or absent"
spasm | 3 months after injury.
  spasm in the injured muscle "present or absent"
Pain with active muscle stretches | 1or 2 days after injury.
  "present or absent"
Pain with active muscle stretches | 2 weeks after injury.
  "present or absent"
Pain with active muscle stretches | 1month after injury.
  "present or absent"
Pain with active muscle stretches | 3 months after injury.
  "present or absent"
Pain with passive muscle stretches | 1 or 2 days after injury.
  "present or absent"
Pain with passive muscle stretches | 2 weeks after injury.
  "present or absent"
pain with passive muscle stretches | 3 months after injury.
  "present or absent"
Pain with passive muscle stretches | 1month after injury.
  "present or absent"
pain with active muscle contraction | 1 or 2 days after injury.
  "present or absent"
pain with active muscle contraction | 2 weeks after injury.
  "present or absent"
pain with active muscle contraction | 1month after injury.
  "present or absent"
pain with active muscle contraction | 3 months after injury.
  "present or absent"
pain with against resistance muscle contraction | 1 or 2 days after injury.
  "present or absent"
pain with against resistance muscle contraction | 2 weeks after injury.
  "present or absent"
pain with against resistance muscle contraction | 1month after injury.
  "present or absent"
pain with against resistance muscle contraction | 3 months after injury.
  "present or absent"
size of injury | 1 or 2 days after injury.
  in cm2 using ultrasound
size of injury | 2 weeks after injury.
  in cm2 using ultrasound
size of injury | 1month after injury.
  in cm2 using ultrasound
size of injury | 3 months after injury.
  in cm2 using ultrasound
disorganized fibrous tissue | 1 or 2 days after injury.
  "present or absent" using ultrasound
disorganized fibrous tissue | 2 weeks after injury.
  "present or absent" using ultrasound
disorganized fibrous tissue | 1month after injury.
  "present or absent" using ultrasound
disorganized fibrous tissue | 3 months after injury.
  "present or absent" using ultrasound
hematoma | 1 or 2 days after injury.
  "present or absent" using ultrasound
hematoma | 2 weeks after injury.
  "present or absent" using ultrasound
hematoma | 1month after injury.
  "present or absent" using ultrasound
hematoma | 3 months after injury.
  "present or absent" using ultrasound
Doppler signal | 1 or 2 days after injury.
  "present or absent" using ultrasound
Doppler signal | 2 weeks after injury.
  "present or absent" using ultrasound
Doppler signal | 1month after injury.
  "present or absent" using ultrasound
Doppler signal | 3 months after injury.
  "present or absent" using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M. Hassanein, Msc, Principal Investigator — Ain Shams University; Wael A.M. Nassar, MD, Study Director — Ain Shams University; Medhat M. Magdy, Msc, Principal Investigator — Ain Shams University; Amr G. Gendya, MD, Principal Investigator — Ain Shams University; Haitham Adel A. A. El Dessokey, MD, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woodhouse JB, McNally EG. Ultrasound of skeletal muscle injury: an update. Semin Ultrasound CT MR. 2011 Apr;32(2):91-100. doi: 10.1053/j.sult.2010.12.002. PMID 21414545